CLINICAL TRIAL: NCT07205068
Title: Improved Outcomes With Pre-Procedure Shockwave IVL of Common Femoral Artery Access Site Prior to Large Bore Access and Pre-Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5319; Institutional Review Board (Other: The University of Tennessee Health Science Center)
Record Dates: First submitted 2025-08-21; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis; Transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Shockwave model (M5) Intravascular Lithotripsy (IVL) (Experimental): Patients will be treated with the Shockwave M5 Intravascular Lithotripsy (IVL) device prior to femoral artery access using the modified Seldinger technique
  Interventions: Device: Shockwave M5 IVL Catheter; Procedure: Modified Seldinger Technique
- Standard femoral access (Active Comparator): Patients will receive standard femoral artery access via the modified Seldinger approach without utilizing intravascular lithotripsy in heavily calcified femoral arteries
  Interventions: Procedure: Modified Seldinger Technique

INTERVENTIONS:
Device: Shockwave M5 IVL Catheter — The Shockwave M5 IVL Catheter is a balloon catheter designed to modify calcified arterial plaque using intravascular lithotripsy prior to vascular access
  Arms: Shockwave model (M5) Intravascular Lithotripsy (IVL)
Procedure: Modified Seldinger Technique — Standard of care for femoral access in patients with calcified femoral arteries
  Arms: Shockwave model (M5) Intravascular Lithotripsy (IVL)
Procedure: Modified Seldinger Technique — Standard femoral artery access using the modified Seldinger technique without any prior vessel preparation or plaque modification.
  Arms: Standard femoral access

SUMMARY:
The primary purpose of this study is to observe reduced access site complications in patients with heavily calcified common femoral arteries requiring Transcatheter Aortic Valve Replacement (TAVR)

DETAILED DESCRIPTION:
This is a prospective randomized/control trial pilot study to compare clinical outcomes of common femoral artery access in patients undergoing TAVR at the University of Tennessee Medical. Specifically, This study compares patients utilizing the Shockwave model (M5) Intravascular Lithotripsy (IVL) prior to standard arterial access using the modified Seldinger technique to those utilizing the standard femoral artery access via the modified Seldinger approach without the utilization of intravascular lithotripsy in heavily calcified femoral arteries.

The secondary purposes of this study are to:

1. Determine the clinical outcomes between groups
2. Distinguish extravasation post closure at the end of the procedure
3. Compare the need for open vascular surgery between groups
4. Examine PTA or Stents to the CFA to help hemostasis or local vascular complications between groups
5. Number of Perclose devices used between groups
6. Compare Bleeding/Hematoma between groups
7. Examine the difference in hospital length of stay between groups
8. Examine renal function post procedure
9. Difference in pain or numbness in the distal extremity between groups
10. Mortality related to complications from vascular closure site between groups
11. Conversion to general anesthesia due to additional procedures required to address the CFA access site complications between groups

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Patient with a diagnosis of severe aortic stenosis undergoing TAVR
3. Participants must be able to read and understand study procedures
4. Willing to participate and sign an ICF
5. Patients with > 90-degree arc of calcium at the large bore access site per CT documentation

Exclusion Criteria:

1. Unable to understand study procedures
2. Unwilling to give consent
3. Patients with cognitive impairments that can affect their ability to give consent
4. Unfavorable calcium distribution of femoral artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-04 (Estimated); Primary Completion 2026-11-04 (Estimated); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate for contrast extravasation post closure of femoral artery at the end of the procedure | Immediately post-procedure

SECONDARY OUTCOMES:
Determine need for Vascular surgery consultation | During hospital stay (Day 0-3)
If vascular complication, was PTA, stenting, or open surgery used | During hospital stay (Day 0-3)
Number of perclose devices used to close the femoral artery access site | During procedure (Day 0)
Determine presence of other vascular complications I.e. bleeding, hematoma, emboli etc | Within 3 days post-procedure
Change in Hemoglobin | Day 0 to Day 3 post-procedure
  As part of evaluating clinical deterioration, this outcome measures the drop in hemoglobin (g/dL)
Change in Serum Creatinine | Day 0 to Day 3 post procedure
  As part of evaluating clinical deterioration, this outcome assesses the increase in serum creatinine (mg/dL)
Incidence of Hypotension or Shock | Day 0 to Day 3 post-procedure
  As part of evaluating clinical deterioration, this outcome captures the number of participants who develop hypotension (SBP < 90 mmHg) or clinical shock.
Incidence of Infections or Sepsis | Day 0 to Day 3 post-procedure
  As part of evaluating clinical deterioration, this outcome records the number of participants diagnosed with infection or sepsis
Determine if there is a difference between hospital length of stay | From date of admission to date of discharge, assessed up to 60 days
  Hospital length of stay will be measured in days from the date of admission to the date of discharge. The total duration will be compared between the intervention and control groups.
Assess for difference in pain/numbness in distal extremities post-procedure (Yes/No) | Within 3 days post-procedure
Assess for differences in mortality related to complications between the groups | Up to 3 months post-procedure
  Presence of new or worsening pain or numbness in the distal extremities will be assessed by patient-reported symptoms during routine clinical evaluation and physical examination. If present, symptoms will be documented in medical records
Failure of treatment | Day 0 to discharge (or up to 3 days post-procedure)
  Failure to achieve the intended procedural outcomes or additional interventions due to complications
Number of related AE(s) | Up to 3 months post-procedure
Number of related SAE(S) | Up to 3 months post-procedure
Side effects reported by subjects or observed by study team | Within 3 days post-procedure, or up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT07205068/Prot_SAP_000.pdf